CLINICAL TRIAL: NCT01448135
Title: Pilot Study Evaluating the Efficacy, Tolerance and Safety of VITAL AF (Semi Elemental, High Protein, High Omega 3 Fat Enteral Formula) Versus Osmolite 1.2 (High Protein Enteral Formula) in Multiple ICU Settings (Medical, Surgical, Cardiothoracic)
Brief Title: Tolerance and Efficacy of a Predigested, High Protein, High Omega 3 Fat Enteral Feeding Formula Versus a Standard Formula In Multiple Intensive Care Unit Settings
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Columbia University (Other)
Collaborators: Abbott Nutrition (Industry)
Responsible Party: Principal Investigator, Ira Jay Goldberg, Dickinson W. Richards, Jr. Professor of Medicine, Columbia University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: AAAI1205; ANUS1015 (Other Grant/Funding Number: ABBOTT Nutrition)
Record Dates: First submitted 2011-10-03; First posted 2011-10-07 (Estimated); Last update posted 2015-06-23 (Estimated); Status verified 2014-01

CONDITIONS: Critical Illness; Enteral Feeding
MeSH Terms: conditions — Critical Illness

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: No

ARMS (2):
- Vital AF (Experimental)
  Interventions: Other: VITAL AF
- Osmolite 1.2 (Active Comparator)
  Interventions: Other: Osmolite 1.2

INTERVENTIONS:
Other: VITAL AF — Semi-elemental, high protein, and high omega-3 fish oil enteral formula
  Arms: Vital AF
Other: Osmolite 1.2 — High protein enteral formula
  Arms: Osmolite 1.2

SUMMARY:
The purpose of this pilot study is to assess the efficacy, safety and tolerance profile of the enteral feeding product VITAL AF (a semi-elemental, high protein, and high omega-3 fish oil) when compared to Osmolite 1.2, a standard feeding product in critically ill and/or post surgical patients in the intensive care unit (ICU). If enough patients are recruited, inferences about impact on outcomes may also be drawn.

ELIGIBILITY:
Inclusion Criteria:

* Subject requires enteral tube feeding as sole source of nourishment
* Subject, or subject's legally acceptable representative (LAR), has provided voluntarily and informed consent form, as deemed appropriate and approved by the Columbia University Medical Center Institutional Review Board
* Subject is ≥ 18 years of age
* Subject is male or non-pregnant female at least six weeks postpartum and non-lactating females of childbearing potential will be required to confirm non-pregnancy status with a pregnancy test at screening
* Subject has an initial APACHE II score less than or equal to 24

Exclusion Criteria:

* Subject requires parenteral nutrition
* Subject is acutely impacted or constipated
* Subject has intestinal obstruction
* Subject is too hemodynamically unstable for enteral feeding
* Subject has an allergy or intolerance to any ingredient in the study product by documentation or verbal report by subject or subject's LAR
* Subject is participating in a non-Abbott approved concomitant trial
* Subject has gastrointestinal disease, including acute pancreatitis, active gastrointestinal bleeding, acute inflammatory bowel disease, or has undergone intestinal surgery within the past month

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2011-10; Primary Completion 2014-11 (Actual); Study Completion 2014-11 (Actual)

PRIMARY OUTCOMES:
Improved tolerance to enteral (tube) feeding | Baseline and 21 Days
  Measure incidence of diarrhea, nausea, vomiting, increased gastric residual, etc.

SECONDARY OUTCOMES:
Improved delivery of prescribed calories | Baseline and 21 Days
  Measurement of volume of feeding product actually delivered to patient is part of the daily flow-sheet data.
Decreased incidence of complications | Baseline and 21 Days
  Measure incidence of diarrhea, nausea, vomiting, increased gastric residual, etc.

CONTACTS AND LOCATIONS:
Overall Officials: Ira J Goldberg, MD, Principal Investigator — Columbia University
Locations (1):
- NewYork-Presbyterian Hospital at Columbia University Medical Center, New York, New York, United States

REFERENCES:
- [Derived] Seres DS, Ippolito PR. Pilot study evaluating the efficacy, tolerance and safety of a peptide-based enteral formula versus a high protein enteral formula in multiple ICU settings (medical, surgical, cardiothoracic). Clin Nutr. 2017 Jun;36(3):706-709. doi: 10.1016/j.clnu.2016.04.016. Epub 2016 Apr 26. PMID 27161892